CLINICAL TRIAL: NCT06900205
Title: Effects of Esketamine on the Incidence of Postoperative Delirium and Postoperative Sleep Disturbance in Elderly Patients After Major Non-cardiac Surgery: A Multi-Center Randomized Controlled Trial
Brief Title: Effects of Esketamine on the Incidence of Postoperative Delirium and Postoperative Sleep Disturbance in Elderly Patients After Major Non-cardiac Surgery
Acronym: EPISODE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial protocol has undergone substantial revisions, including modifications to the primary outcome measure, which fundamentally alter the original study objectives. As these changes are not compatible with the initial registration, we
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Xuhui Central Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-026
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Delirium (POD); Postoperative Sleep Disturbance
Keywords: esketamine; non-cardiac surgery; Postoperative Delirium (POD); Postoperative Sleep Disturbance
MeSH Terms: conditions — Emergence Delirium | interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Drug: Esketamine After anesthesia induction intubation and before surgery,0.25mg/kg esketamine will be diluted into a 10ml syringe and injected intravenously.
  After surgery,a postoperative intravenous analgesia pump will be given with the following drugs and dosages:sufentanil 1.5ug/kg,esketaminge 1.0mg/kg and tolansetron 5mg, diluted into100ml at 2ml/h for 48h.
  Drug: 0.9% saline After anesthesia induction intubation and before surgery,10ml of 0.9% saline will be injected intravenously.
  After surgery,a postoperative intravenous analgesia pump will be given with the following drugs and dosages:sufentanil 1.5ug/kg and tolansetron 5mg, diluted into100ml at 2ml/h for 48h.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- esketamine group (Experimental): The esketamine group patients will be received esketamine perioperatively.
  Interventions: Drug: Esketamine
- Placebo group (Placebo Comparator): The placebo group patients will be received 0.9% saline perioperatively.
  Interventions: Drug: 0.9 % saline

INTERVENTIONS:
Drug: Esketamine — loading dose:intravenous infusion of 0.25mg/kg esketamine after induction of aneshtesia; postoperative intravenous analgesia:1.5ug/kg sufentail+1mg/kg esketamine diluted into 100ml will be provided to the patients after surgery at a rate of 2ml/h for 48h.
  Arms: esketamine group
Drug: 0.9 % saline — loading dose:intravenous infusion the same volume of 0.9% saline as the other group after induction of aneshtesia; postoperative intravenous analgesia:1.5ug/kg sufentail diluted into 100ml will be provided to the patients after surgery at a rate of 2ml/h for 48h.
  Arms: Placebo group

SUMMARY:
Postoperative delirium (POD) is a common surgical complication.It is associated with a range of negative outcomes such as delayed postoperative recovery,prolonged hospitalization,additional medical expenditures and higher mortality.

Meanwhile,sleep disorders are not only an important predisposing factor for delirium,but also one of the main symptoms of delirium.Systemic inflammatory responses caused by sleep disorders may be an important mechanism for POD.

Many studies have shown that esketamie may inhibit inflammatory factors and enhance neuroplasticity.

In summary,we felt the need to further explore the therapeutic potential of esketamine in the area of POD as well as postoperative sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧ 65 years;
2. ASA Ⅰ-Ⅲ;
3. Elective major non-cardiac surgery;
4. Voluntary signed informed consent.

Exclusion Criteria:

1. People with mental illness;
2. Suffering from serious central nervous system disorders such as arkinson's disease, Alzheimer's disease, etc;
3. Elevated intracranial pressure;
4. Emergency or trauma surgery;
5. Prior history of postoperative delirium or postoperative cognitive decline;
6. The patient has impaired hearing or impaired vision;
7. Suffering from severe systemic underlying diseases (e.g. cardiac insufficiency, malignant arrhythmia, malignant hypertension, hepatic failure, renal failure, etc.);
8. The patient is in chronic pain;
9. The patient is severely malnourished;
10. Patients with stage 3 or 4 malignant tumors, pancreatic cancer, allbladder cancer, cholangiocarcinoma and other tumors with high malignancy and poor prognosis.
11. history of allergy to or contraindication to esketamine;
12. inability or unwillingness to complete questionnaires or clinical testing;
13. Unable or unwilling to use a postoperative intravenous analgesic pump.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | postoperative 7 day
  Postoperative delirium is assessed by the 3-minute diagnostic interview for CAM (3D-CAM) or the combination of the Richmond Anxiety Scale (RASS) and the Confusion assessment method for intensive care unit (CAM-ICU) as applicable.
The incidence of postoperative sleep disturbance | postoperative 3 day
  Postoperative sleep disturbance is evaluated by the Athens Insomnia Scale (AIS).
  The AIS is a self-rated psychometric questionnaire to quantify sleep difficulties according to the International Statistical Classification of Diseases and Related Health Problems, Tenth Revision criteria.
  The AIS consists of 8 items: waking up at night, sleep induction, final awakening, total sleep duration, sleep quality, well-being, functional ability, and daytime sleepiness.
  The AIS score ranges from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia.

SECONDARY OUTCOMES:
The incidence of postoperative cognitive dysfunction | 7 days after surgery and 90 days after surgery
  Postoperative delirium is assessed by the Montreal Cognitive Assessment (MoCA).
  MoCA scale was widely identified in the detection of mild cognitive impairment. MoCA assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
  The total possible score is 30 points; a score of 26 or above is considered normal.
postoperative pain severity score | 2 hours after surgery、postoperative 3 day and 90 days after surgery
  The degree of surgical incision pain will be assessed at rest and on movement by Visual Analogue Scale (VAS). VAS ranges from 0 to 10, with the highest score indicating the worst pain.
The incidence of postoperative adverse reactions | postoperative 90 days
  Postoperative adverse reactions within 90 days were defined as postoperative adverse reactions that are new, have an adverse effect on the patient, and require medical intervention (including psychiatric system symptoms, 30-day all-cause mortality etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and de-identified individual participant data could be shared after 1 year after publication with the permission of principle investigator for reasonable usage.
Supporting Information: Study Protocol
Time Frame: The data could be shared after 1 year after publication with the permission of principle investigator. The duration of the data sharing will be determined by principle investigator after publication.
Access Criteria: Study protocol and de-identified individual participant data could be shared after 1 year after publication with the permission of principle investigator. Please email principle investigator if researchers wish to have the data.

REFERENCES:
- [Background] Xiong X, Shao Y, Chen D, Chen B, Lan X, Shi J. Effect of Esketamine on Postoperative Delirium in Patients Undergoing Cardiac Valve Replacement with Cardiopulmonary Bypass: A Randomized Controlled Trial. Anesth Analg. 2024 Oct 1;139(4):743-753. doi: 10.1213/ANE.0000000000006925. Epub 2024 Mar 6. PMID 38446699
- [Background] Luo T, Deng Z, Ren Q, Mu F, Zhang Y, Wang H. Effects of esketamine on postoperative negative emotions and early cognitive disorders in patients undergoing non-cardiac thoracic surgery: A randomized controlled trial. J Clin Anesth. 2024 Aug;95:111447. doi: 10.1016/j.jclinane.2024.111447. Epub 2024 Mar 23. PMID 38522144
- [Background] Zhang A, Zhou Y, Zheng X, Zhou W, Gu Y, Jiang Z, Yao Y, Wei W. Effects of S-ketamine added to patient-controlled analgesia on early postoperative pain and recovery in patients undergoing thoracoscopic lung surgery: A randomized double-blinded controlled trial. J Clin Anesth. 2024 Feb;92:111299. doi: 10.1016/j.jclinane.2023.111299. Epub 2023 Nov 7. PMID 37939610
- [Background] Sadeghirad B, Dodsworth BT, Schmutz Gelsomino N, Goettel N, Spence J, Buchan TA, Crandon HN, Baneshi MR, Pol RA, Brattinga B, Park UJ, Terashima M, Banning LBD, Van Leeuwen BL, Neerland BE, Chuan A, Martinez FT, Van Vugt JLA, Rampersaud YR, Hatakeyama S, Di Stasio E, Milisen K, Van Grootven B, van der Laan L, Thomson Mangnall L, Goodlin SJ, Lungeanu D, Denhaerynck K, Dhakharia V, Sampson EL, Zywiel MG, Falco L, Nguyen AV, Moss SJ, Krewulak KD, Jaworska N, Plotnikoff K, Kotteduwa-Jayawarden S, Sandarage R, Busse JW, Mbuagbaw L. Perioperative Factors Associated With Postoperative Delirium in Patients Undergoing Noncardiac Surgery: An Individual Patient Data Meta-Analysis. JAMA Netw Open. 2023 Oct 2;6(10):e2337239. doi: 10.1001/jamanetworkopen.2023.37239. PMID 37819663
- [Background] Mevorach L, Forookhi A, Farcomeni A, Romagnoli S, Bilotta F. Perioperative risk factors associated with increased incidence of postoperative delirium: systematic review, meta-analysis, and Grading of Recommendations Assessment, Development, and Evaluation system report of clinical literature. Br J Anaesth. 2023 Feb;130(2):e254-e262. doi: 10.1016/j.bja.2022.05.032. Epub 2022 Jul 7. PMID 35810005
- [Background] Sprung J, Roberts RO, Weingarten TN, Nunes Cavalcante A, Knopman DS, Petersen RC, Hanson AC, Schroeder DR, Warner DO. Postoperative delirium in elderly patients is associated with subsequent cognitive impairment. Br J Anaesth. 2017 Aug 1;119(2):316-323. doi: 10.1093/bja/aex130. PMID 28854531
- [Result] Qiu D, Wang XM, Yang JJ, Chen S, Yue CB, Hashimoto K, Yang JJ. Effect of Intraoperative Esketamine Infusion on Postoperative Sleep Disturbance After Gynecological Laparoscopy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2244514. doi: 10.1001/jamanetworkopen.2022.44514. PMID 36454569
- [Result] Avidan MS, Maybrier HR, Abdallah AB, Jacobsohn E, Vlisides PE, Pryor KO, Veselis RA, Grocott HP, Emmert DA, Rogers EM, Downey RJ, Yulico H, Noh GJ, Lee YH, Waszynski CM, Arya VK, Pagel PS, Hudetz JA, Muench MR, Fritz BA, Waberski W, Inouye SK, Mashour GA; PODCAST Research Group. Intraoperative ketamine for prevention of postoperative delirium or pain after major surgery in older adults: an international, multicentre, double-blind, randomised clinical trial. Lancet. 2017 Jul 15;390(10091):267-275. doi: 10.1016/S0140-6736(17)31467-8. Epub 2017 May 30. PMID 28576285